CLINICAL TRIAL: NCT05961553
Title: Effect of an Individual Counseling Session on Physical Activity Level of Individuals With Chronic Obstructive Pulmonary Disease (COPD) - Randomized Controlled Study (RCT)
Brief Title: Effect of an Individual Counseling Session on Physical Activity Level of Individuals With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polytechnic Institute of Porto (Other)
Responsible Party: Principal Investigator, Tiago Miguel dos Santos Pastilha, Principal Investigator, Polytechnic Institute of Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16.OBS.2020
Record Dates: First submitted 2023-07-16; First posted 2023-07-27 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: COPD
Keywords: COPD; Pulmonary Rehabilitation; Physical Activity; Counseiling Session; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity Counseling + Pulmonary Rehabilitation (Experimental): The counseling session on physical activity was carried out individually, six weeks after starting the respiratory rehabilitation program, with an average duration of 30 minutes, based on the guidelines of the Living Well with COPD program. The main objective of the session was: to help the participant and family members to increase physical activity levels and their integration in the long term and as secondary objectives; reinforce the importance and benefits of physical activity in the management of the health condition/symptoms; plan daily/weekly moments of physical activity; define daily goals (physical activity time/sitting time) attainable for each participant; integrate family members/companions into the user's physical activity plan; clarify doubts of the user/relative about the theme.
  Interventions: Behavioral: Physical Activity Counseling session; Other: Pulmonary Reabilitation
- Pulmonary Rehabilitation (Active Comparator): The program comprises a hospital group exercise program, twice a week, on alternate days, for 1h30 to 2h, each session, which included: monitoring of vital signs, peripheral oxygen saturation (SpO2), subjective perception of exertion (RPE), dyspnea and body mass; warm-up phase (10min), with ventilatory control and low-intensity upper and lower limb exercises; continuous aerobic training phase, performed on a treadmill, static cycle ergometer and/or arm ergometer (30-45min), at 60-80% of the maximum Cardiopulmonary Exercise Test load; strength training phase, with free weights, machines (10-20min), at 50-80% of the Maximum Repetition (RM), (8-12 repetitions), 1-2 sets, 8-10 exercises ( upper limbs, trunk and lower limbs); cooling phase (5-10min), with 5 to 8 relaxation, stretching and ventilatory control exercises. The progression of training loads is carried out according to RPE and dyspnea, safeguarding SpO2 values above 88-90% and Heart Rate below the maximum defined for training.
  Interventions: Other: Pulmonary Reabilitation

INTERVENTIONS:
Behavioral: Physical Activity Counseling session — The counseling session on physical activity was carried out individually, six weeks after starting the respiratory rehabilitation program, with an average duration of 30 minutes, based on the guidelines of the Living Well with COPD program. The main objective of the session was: to help the participant and family members to increase physical activity levels and their integration in the long term and as secondary objectives; reinforce the importance and benefits of physical activity in the management of the health condition/symptoms; plan daily/weekly moments of physical activity; define daily goals (physical activity time/sitting time) attainable for each participant; integrate family members/companions into the user's physical activity plan; clarify doubts of the user/relative about the theme.
  Arms: Physical Activity Counseling + Pulmonary Rehabilitation
Other: Pulmonary Reabilitation — The program comprises a hospital group exercise program, twice a week, on alternate days, for 1h30 to 2h, each session.

SUMMARY:
The goal of this randomized clinical trial is to study the effect of an individual counseling session on the level of physical activity and motivation to practice physical exercise in individuals with COPD. The main question[s] it aims to answer are:

• Does a counseling session improve the level of physical activity and motivation to practice physical exercise in individuals with COPD?

Participants will perform a respiratory rehabilitation program (Control Group, CG) and a respiratory rehabilitation program and the counseling session (Experimental Group, EG).

Researchers will compare EG to CG to see if there is any difference in physical activity level and motivation to exercise between groups.

ELIGIBILITY:
Inclusion Criteria:

* Portuguese nationality;
* Medical diagnosis of COPD according to Global Initiative for Chronic Obstructive Lung Disease (GOLD 2022);
* Aged over 40 years.

Exclusion Criteria:

* underwent recent orthopedic surgeries (<3 months);
* Pregnant;
* Terminal illness diagnosis (life expectancy of less than 6 months);
* High cardiovascular risk classification for the practice of physical activity according to American College of Sports Medicine (ACSM 2018).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Average Daily Steps | 7 days
  quantitative variable met through the daily average of the steps, using accelerometer data.
Light Physical Activity | 7 days
  quantitative variable evaluated with the accelerometer, measured in minutes.
Moderate Physical Activity | 7 days
  quantitative variable evaluated with the accelerometer, measured in minutes.
Vigorous Physical Activity | 7 days
  quantitative variable evaluated with the accelerometer, measured in minutes.
Sedentary Activity | 7 days
  quantitative variable evaluated with the accelerometer, measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Tiago Pastilha, PT, Principal Investigator — Escola Superior de Saúde; Ana Alexandrino, PhD, Study Director — Escola Superior de Saúde; Susana Vale, PhD, Study Director — Escola Superior de Educação; Rui Macedo, PhD, Study Director — Escola Superior de Saúde
Locations (1):
- Hospital Distrital da Figueira da Foz, EPE, Figueira da Foz Municipality, Coimbra District, Portugal

IPD SHARING:
Plan to Share IPD: No